CLINICAL TRIAL: NCT01070173
Title: Ghrelin Levels in Children With Gastrointestinal Symptoms and/or Poor Growth
Brief Title: Ghrelin Levels in Children With Poor Growth
Status: Completed | Type: Observational
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jordan Pinsker, Chief, Pediatric Endocrinology, Tripler Army Medical Center
Other Study IDs: 5H08
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-01

CONDITIONS: Idiopathic Short Stature; Failure to Thrive
Keywords: Ghrelin; short stature; failure to thrive
MeSH Terms: conditions — Failure to Thrive; Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Short Stature: Poor linear growth
- Poor Weight Gain (Failure-To-Thrive): Poor Weight Gain
- Isolated Gastrointestinal Symptoms: No growth symptoms

SUMMARY:
The investigators hypothesize that low serum ghrelin levels may characterize a group of patients with poor weight gain and/or linear growth who do not have any other identified cause for growth failure. These patients may present with a variety of complaints and are often evaluated by both pediatric endocrinologists and pediatric gastroenterologists. The investigators hypothesize that ghrelin has a physiologically important role in linear growth and that chronic diseases of the gastrointestinal system, such as H. Pylori infection or celiac disease, may alter serum ghrelin levels in children. Low ghrelin levels may be a factor leading to poor growth, potentially by altering growth hormone secretion and/or by decreasing appetite. By measuring ghrelin levels in children with short stature and in children with gastrointestinal disease, the investigators will further elucidate the possible physiologic role of ghrelin in childhood growth and how it may be altered in conditions causing short stature and in certain gastrointestinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the short stature group, subjects must have had short stature, defined height less than -2 SD for gender and age or an abnormal growth velocity for gender and age).
* To be included in the failure-to-thrive group, subjects must have had poor weight gain, defined as weight less than -2 SD for gender and age or an abnormal weight velocity for gender and age.
* Patients in both groups will be evaluated for the presence of chronic gastrointestinal symptoms, defined as symptoms of gastrointestinal disease for greater than 6 weeks or recurrent symptoms. Patients who were affected in both weight and height will be stratified by which measurement was more severely affected, with poor weight gain being the primary problem in the "failure-to-thrive" grouping (Group 2) and "poor linear growth" being the primary problem in the short stature group (Group 1).
* Patients who have had chronic gastrointestinal symptoms, defined as symptoms of gastrointestinal disease for greater than 6 weeks or recurrent symptoms, but normal stature and growth, will be analyzed separately (Group 3).

Exclusion Criteria:

* Must not have a known diagnosis as an etiology for growth failure or GI symptoms prior to presentation.

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Twenty-five (25) patients seen for evaluation of short stature in the pediatric endocrinology clinic will have serum ghrelin levels measured in addition to their usual routine bloods tests.
  Twenty-five (25) patients will be selected from patients who present with chronic gastrointestinal symptoms (symptoms of gastrointestinal disease for greater than 6 weeks or recurrent symptoms) and who have poor growth.
  The remaining 25 will be selected from patients with chronic gastrointestinal symptoms (symptoms of gastrointestinal disease for greater than 6 weeks or recurrent symptoms) who have normal growth.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Principal Investigator — Tripler Army Medical Center
Locations (1):
- Tripler Army Medical Center/Dept of Pediatrics, Tripler AMC, Hawaii, United States

REFERENCES:
- [Result] Pinsker JE, Ondrasik D, Chan D, Fredericks GJ, Tabisola-Nuesca E, Fernandez-Aponte M, Focht DR, Poth M. Total and acylated ghrelin levels in children with poor growth. Pediatr Res. 2011 Jun;69(6):517-21. doi: 10.1203/PDR.0b013e3182181b2c. PMID 21386753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-two patients were recruited into the study.
Groups:
- Short Stature: Poor linear growth Group
- Poor Weight Gain (Failure-To-Thrive): Poor Weight Gain (Failure-To-Thrive) Group
- Isolated Gastrointestinal Symptoms: Isolated Gastrointestinal Symptoms Group
Period: Overall Study
Arm/Group | Short Stature | Poor Weight Gain (Failure-To-Thrive) | Isolated Gastrointestinal Symptoms
Started | 33 | 8 | 11
Completed | 33 | 8 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Poor Weight Gain (Failure-To-Thrive): Poor Weight Gain (Failure-To-Thrive)
- Isolated Gastrointestinal Symptoms: Isolated Gastrointestinal Symptoms
- Total: Total of all reporting groups
Arm/Group | Short Stature | Poor Weight Gain (Failure-To-Thrive) | Isolated Gastrointestinal Symptoms | Total
Number analyzed (Participants) | 33 | 8 | 11 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 8 | 11 | 52
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 4 | 22
  Male | 19 | 4 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Total Ghrelin Level
Time Frame: Will be measured with baseline screening labs at enrollment.
Population: All participants.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Short Stature | Poor Weight Gain (Failure-To-Thrive) | Isolated Gastrointestinal Symptoms
Number analyzed (Participants) | 33 | 8 | 11
pg/mL | 1063 (77) | 1264 (245) | 1157 (105)

2. Primary Outcome: Acylated Ghrelin Level
Time Frame: Will be measured with baseline screening labs at enrollment.
Population: All participants.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Short Stature | Poor Weight Gain (Failure-To-Thrive) | Isolated Gastrointestinal Symptoms
Number analyzed (Participants) | 33 | 8 | 11
pg/mL | 190 (34) | 465 (128) | 176 (37)

ADVERSE EVENTS:
Arm/Group | Short Stature | Poor Weight Gain (Failure-To-Thrive) | Isolated Gastrointestinal Symptoms
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/33 | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No